CLINICAL TRIAL: NCT03955666
Title: PREVAIL 1: A Phase 1b, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of PRV-3279 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of PRV-3279 in Healthy Subjects
Acronym: PREVAIL1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Provention Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRV-3279-1b
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2019-12

CONDITIONS: Safety

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, multiple ascending dose study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (PRV-3279 or placebo) (Experimental): Sterile solution for intravenous administration, 3 doses, every 2 weeks
  Interventions: Biological: PRV-3279 or placebo
- Cohort B (PRV-3279 or placebo) (Experimental): Sterile solution for intravenous administration, 3 doses, every 2 weeks
  Interventions: Biological: PRV-3279 or placebo

INTERVENTIONS:
Biological: PRV-3279 or placebo — bi-specific antibody-based molecule

SUMMARY:
This Phase 1b study will evaluate the safety of PRV-3279 in healthy adult subjects

DETAILED DESCRIPTION:
PRV-3279-1b is a Phase 1b, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of PRV-3279 in Healthy Subjects.

Eligible subjects include healthy male or female adults, 18 to 50 years of age. Each subject will receive the assigned treatment over 29 days followed by a 56-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations.
2. Body mass index (BMI) 18 to 32 kg/m2, inclusive.
3. Male or female 18 to 50 years of age, inclusive.
4. Nonpregnant women of childbearing potential (WOCBP) and sexually active men must agree to use effective birth control with male contraception during study participation through at least 3 months after the final dose. Women of non-childbearing potential may participate.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Evidence of active or chronic infections.
3. Previous exposure to PRV-3279.
4. Any reason that, in the opinion of the Investigator, would contraindicate the subject's participation in the study or confound the results of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | 85 days
  Assessment of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Provention Bio, Inc.
Locations (1):
- Clinical site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No